CLINICAL TRIAL: NCT07320924
Title: Patient-specific Reconstruction Plate for Alloplastic Bridging of Segmental Mandibular Defects. A Clinical and Radiographic Study.
Brief Title: Patient-specific Reconstruction Plate for Segmental Mandibular Defects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-12-25/PSRP
Record Dates: First submitted 2025-12-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Mandibular Resection; Mandibular Reconstruction* / Methods; Mandibular Reconstruction
Keywords: mandibular resection; surgery; computer-assisted; computer-aided design; computer-aided manufacturing; software

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient specific reconstruction plate (Experimental): patient with mandibular ablation defect managed with patient specific reconstruction plate
  Interventions: Device: Patient specific reconstruction plate

INTERVENTIONS:
Device: Patient specific reconstruction plate — Patient specific reconstruction plate

SUMMARY:
The mandible's horseshoe-shaped anatomy makes the reconstruction of segmental defects a challenging procedure. Conventional reconstruction typically relies on alloplastic plates to bridge bony stumps; however, these require extensive intraoperative bending, often resulting in imperfect adaptation, press-to-contact fixation, and residual stresses that increase the risk of hardware fatigue and fracture. Recent advances in computer-aided design and manufacturing (CAD/CAM) and virtual surgical planning (VSP) have improved precision in maxillofacial reconstruction. Patient-Specific Reconstruction Plates (PSRP), developed from virtual planning and patient-specific anatomical data, offer a bespoke contour adaptation, predictable screw positioning, and elimination of press-fit deformation. This customization improves alignment, mechanical stability, and long-term outcomes.

DETAILED DESCRIPTION:
The study aims to assess the clinical performance and morbidity rate of computer-guided PSRP in the management of mandibular segmental defects.

This prospective interventional clinical trial will be conducted on a total of 14 patients with a segmental mandibular defect, recruited from Alexandria University Teaching Hospital. All patients will be reconstructed using a PSRP alloplastic bridging plate, utilizing a preoperative virtual surgical planning and design. Patients will be evaluated clinically for the rate of morbidity and range of mandibular excursions. Furthermore, postoperative radiographic 3D analysis will evaluate the accuracy of the computer-guided procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a segmental mandibular continuity defect, not involving the condyle.
2. Patients suffering from benign, locally invasive or malignant lesions that involving the lower border of the mandible.
3. Patients with recurrent lesions after resection.
4. Patients dealing with osteomyelitis or jaw osteonecrosis that is indicated for sequestrectomy.

   • Stage-III jaw osteonecrosis.
5. Patients with traumatic defects.
6. Patients with post-gunshot mandibular defects.

Exclusion Criteria:

1. Medically compromised patients contradict the operation.
2. Patients with segmental mandibular defects that require condylar process resection
3. Patients with lateral segmental mandibular defects involving the condyle that require reconstruction using an alloplastic total joint.
4. Patients with an active infection at the site of resection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications and degree of morbidity | 3 months
  All patients will be assessed immediately post-operative, at 1 and 3 months. Any complication that arises during the clinical follow-up period will be monitored and reported. Complications include prolonged hospital stay, prolonged drug administration, signs of screw or PSRP loosening, PSRP fracture, wound dehiscence or tissue necrosis, Intra/extraoral PSRP exposure, and fistulae.

SECONDARY OUTCOMES:
Functional Range of Mandibular Excursions | 3 months
  The range of mandibular excursions will be objectively recorded using a caliper measurement during the clinical follow-up periods. The following excursions will be recorded:
  Intra-Incisal Mouth Opening (I-IMO) Dental Midline Deflection on Opening (DMD-O) Chin Midline Deflection on Opening (CMD-O)

CONTACTS AND LOCATIONS:
Overall Officials: yehia M El-Mahallawy, Phd, Principal Investigator — Faculty of Dentistry, Alexandria University, Alexandria, Alexandria
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
All data will be de-identified to protect the participant data. patients signed an informed consent for the use of their medical records and data for study.